CLINICAL TRIAL: NCT04321356
Title: Analysis of Competitive PCR and PS Total Knee Arthroplasty
Brief Title: Analysis of Competitive Posterior Cruciate Retaining (PCR) and Posterior Stabilized (PS) Total Knee Arthroplasty (TKA)
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Richard Komistek, Principal Investigator, The University of Tennessee, Knoxville
Other Study IDs: 3187FB WIRB20180745 Extension
Record Dates: First submitted 2019-12-19; First posted 2020-03-25 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-02

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty; Knee
Keywords: Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (4):
- Stryker Triathlon PCR TKA: Subjects implanted with a Stryker Triathlon PCR TKA
  Interventions: Device: Triathlon PCR TKA
- Stryker Triathlon PS TKA: Subjects implanted with a Stryker Triathlon PS TKA
  Interventions: Device: Triathlon PS TKA
- Zimmer Persona PCR TKA: Subjects implanted with a Zimmer Persona PCR TKA
  Interventions: Device: Persona PCR TKA
- Zimmer Persona PS TKA: Subjects implanted with a Zimmer Persona PS TKA
  Interventions: Device: Persona PS TKA

INTERVENTIONS:
Device: Triathlon PCR TKA — Total Knee Arthroplasty System
  Groups: Stryker Triathlon PCR TKA
Device: Triathlon PS TKA — Total Knee Arthroplasty System
  Groups: Stryker Triathlon PS TKA
Device: Persona PCR TKA — Total Knee Arthroplasty System
  Groups: Zimmer Persona PCR TKA
Device: Persona PS TKA — Total Knee Arthroplasty System
  Groups: Zimmer Persona PS TKA

SUMMARY:
The purpose of the study is to acquire kinematic in vivo fluoroscopy data from subjects who were implanted with Stryker Posterior Cruciate Retaining (PCR) , Stryker Posterior Stabilized (PS), Zimmer PCR, and Zimmer PS Total Knee Arthroplasty (TKAs). Our lab has previously collected data for the Smith & Nephew PCR, bi-cruciate retaining (BCR), and bi-cruciate stabilized (BCS) TKA.

DETAILED DESCRIPTION:
The objective for this study is to analyze the in vivo kinematics for subjects implanted with either a Stryker PCR, Stryker PS, Zimmer PCR, and Zimmer PS TKA and to compare those patterns to subjects having a normal knee from our previous study and to those patterns from subjects having a Smith & Nephew PCR, BCR, and BCS TKA.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will have one of the following implant types: 1) Stryker Triathlon PCR TKA (28 subjects), 2) Stryker Triathlon PS TKA (28 subjects), 3) Zimmer Persona PCR TKA (28 subjects) and 4) Zimmer Persona PS TKA (28 subjects).
2. Patients must be at least three months post-operative.
3. Participants must not experience any pain or other post-operative complications.
4. Participants must have a stable TKA and be capable of performing a deep knee bend activity.
5. Participants must weigh less than 300 lbs., not underweight (BMI < 18.5) or too obese (BMI>35).
6. Must be in the age range of 18 years to 85 years (both inclusive).
7. Participants must be able to perform the required activities without concern.
8. Subjects must be willing to sign the Informed Consent (IC) form to participate in the study.
9. Patients who do not have previous surgery on the implanted knee that might restrict their movement.

Exclusion Criteria:

1. Pregnant, potentially pregnant, lactating females or of childbearing age. To satisfy radiation protocol, each female subject will be asked if she is pregnant, or possibly could be pregnant. A pregnant person will not be allowed to participate in the study. (All potential female study patients will be asked if they are premenopausal or if they have undergone a hysterectomy. If the possibility of pregnancy exists, a pregnancy kit will be given to the patient at the informed consent meeting, just prior to the fluoro. Results of the test will be recorded in a test log. Any female patient showing a positive test will be excluded from testing.)
2. Subjects without the required type of knee implant.
3. Cannot have pain in other parts of the body that would prohibit the subject from performing the activities).
4. Cannot have ligamentous pain and/or laxity.
5. Unwilling to sign IC/HIPAA form(s).
6. Does not speak English.
7. Patients who have enrolled in a fluoroscopic kinematic study within the past year.
8. Patients currently involved in any personal injury litigation, medical/legal or worker's compensation claims.
9. Patients with known drug or alcohol abuse histories or psychological disorders that could affect ability to complete all aspects of the study.
10. Patients with neurological or musculoskeletal disorders that might adversely affect weight-bearing motion ability.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with a Stryker Triathlon PCR, Stryker Triathlon PS, Zimmer Persona PCR, or Zimmer Persona PS total knee arthroplasty (TKA) implanted by Dr. Harold E. Cates.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Komistek, PhD, Principal Investigator — The University of Tennessee
Locations (2):
- United States (2):
  - Tennessee Orthopaedic Clinic, Knoxville, Tennessee
  - The University of Tennessee, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Researchers would like to retain this study data in our secure database so as to continue to add relevant, current data to our digital collection to help us work with manufacturers in the future to create better implants that last longer and will not require revision surgery. Participants will be asked if their study data may remain a part of the University of Tennessee's Center for Musculoskeletal Research data collection for use in future studies in the IC. Identifiers are automatically removed from the database upon entry into the secure server. Data shared with sponsors is de-identified.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stryker Triathlon PCR TKA | Stryker Triathlon PS TKA | Zimmer Persona PCR TKA | Zimmer Persona PS TKA
Started | 31 | 26 | 29 | 14
Completed | 31 | 26 | 29 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stryker Triathlon PCR TKA | Stryker Triathlon PS TKA | Zimmer Persona PCR TKA | Zimmer Persona PS TKA | Total
Number analyzed (Participants) | 31 | 26 | 29 | 14 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 26 | 29 | 14 | 100
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 17 | 8 | 49
  Male | 19 | 14 | 12 | 6 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31 | 26 | 29 | 14 | 100

OUTCOME MEASURES:

1. Primary Outcome: Medial AP Translations, in mm, During Deep Knee Bend (DKB) Activity
Description: Anterior Posterior (AP) translations, in mm, of medial femoral condyle during deep knee bend activity. Positive values indicate anterior motion of the medial femoral condyle, and negative values indicate posterior motion of the medial femoral condyle.
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Stryker Triathlon PCR TKA | Stryker Triathlon PS TKA | Zimmer Persona PCR TKA | Zimmer Persona PS TKA
Number analyzed (Participants) | 31 | 26 | 29 | 14
millimeters | 4.2 (3.6) | -0.4 (3.4) | -0.5 (2.1) | -3.3 (4.8)

2. Primary Outcome: Lateral AP Translations, in mm, During Deep Knee Bend (DKB) Activity
Description: Anterior Posterior (AP) translations, in mm, of lateral femoral condyle during deep knee bend activity. Positive values indicate anterior motion of the lateral femoral condyle, and negative values indicate posterior motion of the lateral femoral condyle.
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Stryker Triathlon PCR TKA | Stryker Triathlon PS TKA | Zimmer Persona PCR TKA | Zimmer Persona PS TKA
Number analyzed (Participants) | 31 | 26 | 29 | 14
millimeters | 0.7 (3.6) | -3.3 (3.5) | 0.6 (2.3) | -5.2 (4.8)

3. Primary Outcome: Maximum Flexion, in Degrees, During Deep Knee Bend Activity
Description: Maximum weight-bearing flexion, in degrees, during deep knee bend activity
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Stryker Triathlon PCR TKA | Stryker Triathlon PS TKA | Zimmer Persona PCR TKA | Zimmer Persona PS TKA
Number analyzed (Participants) | 31 | 26 | 29 | 14
degrees | 107 (11) | 101 (16) | 107 (11) | 114 (17)

4. Primary Outcome: Axial Rotation, in Degrees, During Deep Knee Bend Activity
Description: Axial rotation (AR), in degrees, during deep knee bend activity. Positive values indicate external femorotibial axial rotation, and negative values indicate internal femorotibial axial rotation.
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Stryker Triathlon PCR TKA | Stryker Triathlon PS TKA | Zimmer Persona PCR TKA | Zimmer Persona PS TKA
Number analyzed (Participants) | 31 | 26 | 29 | 14
degrees | 4.3 (4.4) | 3.6 (3.7) | -1.5 (4.0) | 2.8 (4.7)

ADVERSE EVENTS:
Time Frame: Adverse events would occur and therefore are collected only during the single day of data collection. Thus, we would know right away, and therefore the specific time period is 1 day. There is no participant follow up after data collection, and participants were not monitored after data collection.
Arm/Group | Stryker Triathlon PCR TKA | Stryker Triathlon PS TKA | Zimmer Persona PCR TKA | Zimmer Persona PS TKA
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/26 | 0/29 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/26 | 0/29 | 0/14
Other Adverse Events (participants affected / at risk) | 0/31 | 0/26 | 0/29 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT04321356/Prot_SAP_000.pdf